CLINICAL TRIAL: NCT06926309
Title: THE EFFECT OF PEER MENTORING ON THE KNOWLEDGE, SKILLS, AND METACOGNITIVE THINKING SKILLS OF NURSING STUDENTS ON POSTPARTUM PERINEAL CARE: AN EXPERIMENTAL TRIAL WITH ONE-GROUP PRETEST-POSTTEST DESIGN
Acronym: Perineal care
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Olga Incesu, PhD, Istanbul University - Cerrahpasa
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Florence Nightingale Faculty-4
Record Dates: First submitted 2025-03-18; First posted 2025-04-13 (Actual); Last update posted 2025-04-13 (Actual); Status verified 2025-04

CONDITIONS: Postpartum Perineal Care; Peer Mentoring
Keywords: peer mentoring, skill, postpartum perineal care, undergraduate nursing student, metacognitive thinking

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Experimental (Experimental): Postpartum perineal care training will be given to the experimental group through peer mentoring. The training will last 4 hours in total.
  Interventions: Other: Peer mentoring

INTERVENTIONS:
Other: Peer mentoring — The peer mentor selected by the researchers will be given postpartum perineal care education and peer mentoring education. The peer mentor will prepare perineal care education materials under the supervision of the researchers. Then, the experimental group will be divided into small groups and given 4 hours of perineal care education to their peers.

SUMMARY:
Postpartum perineal care (PPC) is one of the critical skills that should be acquired by students studying in Obstetrics and Gynaecology Nursing under nursing education. Perineal care is a skill that contributes positively to the recovery process of the mother by eliminating the risk of infection through maintaining hygiene of the sutured or non-sutured perineum in postpartum women Peer mentoring is important for both the peer mentor and the peer to practice in accordance with PPC protocols by going through a bidirectional learning experience, for these practices to be evaluated by peer mentors, and for the skill to be experienced in a safe environment. Peer mentoring plays an important role in teaching metacognitive thinking skills as well as the knowledge and skills of peers in nursing education. Although there are studies on the acquisition of skills in peer mentoring in the literature, no study has been found to demonstrate the effect of peer mentoring on the PPC knowledge, skills and metacognitive thinking skills of nursing students. In this context, it is thought that the study will contribute to the literature.

DETAILED DESCRIPTION:
Peer mentoring is one of the methods that emphasises learning as a social process and supports the learning process by sharing knowledge and experience with their/similar (in terms of age, gender, educational background, social status, etc.) peers (Gazula et al., 2017; Sancı & Kelleci, 2019). Peer mentoring is an important process that reinforces and supports learning among peers on personal, social and academic issues (Gazula et al., 2017; Motsaanaka, Makhene & Ally, 2020; Şenyuva & Akince Kocaağalar, 2020).

Peer mentoring in nursing education is important for both reinforcing theoretical knowledge and supporting learning from each other by improving skills during practice (Motsaanaka, Makhene & Ally, 2020; Sözer, 2022). During this process, more experienced nursing students (peer mentors) guide less experienced nursing students (peers), share their professional knowledge, and transfer their experiences. Moreover, peers practice skills with peer mentors and exchange ideas (Gray et al., 2019; Sundlera et al., 2019; Şenyuva & Akince Kocaağalar, 2020). Pinks et al., (2021) have found that peer mentoring facilitates the learning processes of students, improves their skills in problem-solving, learning how to learn, interpersonal communication and empathy, and promotes emotional expression and coping skills focused on emotions (Pinks et al., 2021). Different studies have also emphasised the importance of peer mentoring in acquiring academic and individual adjustment, professional motivation, social-emotional learning and clinical skills. Moreover, it has been shown that students experience adjustment problems when they get into the university and receive support from their peer mentors on issues such as regulations, communication with tutors, school activities and study (Aslan & Erci, 2021; Aydemir, 2024; Bahar, Kocaçal & Maraş, 2022; Fard et al., 2020; Korkut & Başer, 2023; Pehlivan Coştu & Bilgiç, 2023; Shohani et al., 2020; Sözer, 2022).

Peer mentoring eliminates the hierarchical relationship and power imbalance between tutors and students (Ko, Issenberg & Roh, 2022; Şenyuva & Akince Kocaağalar, 2020). Peer mentoring is utilised in nursing education to provide nursing students with knowledge and attitudes as well as psychomotor skills education (Arasteh, Ghezeljeh, & Haghani, 2018; Aslan & Erci, 2021; Bahar, Kocaçal & Maraş, 2022; Carey et al., 2019; Cheraghi et al., 2021; Dikmen ve ark., 2017; Fard et al., 2020; Kim, 2020; Korkut & Başer, 2023; Öztürk, Aközlü & Taşdelen, 2023; Pålsson et al., 2017; Pehlivan Coştu & Bilgiç, 2023; Shohani et al., 2020; Kim, 2020).

The postpartum period is a time when the mother and the baby need much nursing care. The nursing care to be provided during this period is crucial to support both the mother, the newborn and the family to meet their needs. The postpartum period covers the post-natal recovery process of the mother and perineal care is critical for the prevention of infections during this period. The Postpartum Care Management Guide stresses that perineal care is an important practice during the postpartum period (Şimşek & Esencan, 2017). Postpartum perineal care (PPC) is one of the critical skills that should be acquired by students studying in Obstetrics and Gynaecology Nursing under nursing education. Perineal care is a skill that contributes positively to the recovery process of the mother by eliminating the risk of infection through maintaining hygiene of the sutured or non-sutured perineum in postpartum women (Demirci et al., 2014; Şimşek & Esencan, 2017). Peer mentoring is important for both the peer mentor and the peer to practice in accordance with PPC protocols by going through a bidirectional learning experience, for these practices to be evaluated by peer mentors, and for the skill to be experienced in a safe environment (Aslan & Erci, 2021).

Peer mentoring plays an important role in teaching metacognitive thinking skills as well as the knowledge and skills of peers in nursing education (Hattie & Timperley, 2007; Topping, 2009). Metacognition refers to the student's awareness of own thinking processes and his/her ability to control/manage these processes. It is an element that supports the student in gaining the ability to learn on their own. It involves critical, logical, reflective, metacognitive and creative thinking and becomes active when facing problems, uncertainties, questions or dilemmas (Karaoğlan-Yılmaz et al., 2019). While peer mentoring teaches PPC knowledge and skills, discussions between peer mentors and peers raise awareness of metacognitive processes. Feedback from peer mentors helps peers recognise their mistakes and critically evaluate and organise their own thinking processes. It allows them to develop their cognitive process skills by observing their thinking and problem-solving strategies. This allows peers who get peer mentoring to improve their problem-solving skills and offer more effective solutions to the problems they face/will face in clinical settings during perineal care, practice perineal care skills independently, and become competent in skills such as critical decision-making, critical thinking, analytical thinking (Motsaanaka, Makhene & Ally, 2020; Joung et al., 2020; Pinks et al., 2021).

Although there are studies on the acquisition of skills in peer mentoring in the literature, no study has been found to demonstrate the effect of peer mentoring on the PPC knowledge, skills and metacognitive thinking skills of nursing students. In this context, it is thought that the study will contribute to the literature.

ELIGIBILITY:
Inclusion Criteria:receiving no training on postpartum perineal care before, not working part/full-time employment as a nurse -

Exclusion Criteria:Not having given written and verbal consent to participate in the study

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-03-20 (Actual); Primary Completion 2025-05-22 (Estimated); Study Completion 2025-06-28 (Estimated)

PRIMARY OUTCOMES:
Metacognitive Thinking Skills Scale | 2 weeks post intervention
  Metacognitive Thinking Skills Scale of the intervention group change after web based education
Postpartum Perineal Care Skill and Knowledge | 2 weeks post intervention
  Skill and Knowledge of Postpartum Perineal Care point of the intervention group change after web based education

CONTACTS AND LOCATIONS:
Locations (1):
- Florence Nightingale Faculty of Nursing, Istanbul, Şişli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No